CLINICAL TRIAL: NCT06787417
Title: Kinematic and Mechanical Alignment Randomized Trial (KMART): A Technology-Focused Randomized Controlled Trial
Brief Title: Kinematic and Mechanical Alignment Randomized Trial
Acronym: KMART
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Research Institute of St. Joseph's Hamilton (Unknown); Canadian Orthopaedic Foundation (funding) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMART
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
Keywords: Total Knee Arthroplasty; Kinematic Alignment; Mechanical Alignment; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Alignment (Active Comparator)
  Interventions: Procedure: Mechanically-Aligned Arthroplasty
- Restricted Kinematic Alignment (Experimental)
  Interventions: Procedure: Restricted Kinematically-aligned Arthroplasty

INTERVENTIONS:
Procedure: Restricted Kinematically-aligned Arthroplasty — Robot Assisted with Restricted Kinematically-Aligned TKA.
  Arms: Restricted Kinematic Alignment
Procedure: Mechanically-Aligned Arthroplasty — Robot Assisted with Mechanically Aligned TKA.
  Arms: Mechanical Alignment

SUMMARY:
Knee replacement surgery is the second most common surgery in Canada. People who have very painful knee arthritis usually receive a knee replacement where the surgeon aims to make everyone's knee as straight as possible (called mechanical alignment). Mechanical alignment focuses on making the implant last as long as possible. However, everybody's knee shape is different and we think that it is important to take individual differences into account. A newer technique that is more personalized is called restricted kinematic alignment. This technique customizes the placement of the new knee to reproduce each patient's unique knee shape, which may not be perfectly straight. We think this newer technique may feel more natural, be more stable, and lead to better knee function. Restricted kinematic alignment might last as long or longer than mechanical alignment, but the research that has been conducted to date is not clear. We are conducting this study to help surgeons better understand which technique is better. One of the reasons the existing research is not clear is because new developments in robotic technology now allow surgeons to place knee implants very precisely, which was not done in most previous research. In this study everyone will receive a robot-assisted knee surgery so we can be sure the implants are placed as precisely as possible.

The purpose of this trial is to determine whether there are differences in patient outcomes using restricted kinematic alignment rather than the traditionally used mechanical alignment for total knee replacements.

Participants who are having total knee replacements will be randomized to receive either a robot-assisted total knee replacement using mechanical alignment, or a robot-assisted total knee replacement using restricted kinematic alignment . We will ask participants to walk in a markerless motion capture system which will measure walking characteristics at pre-op, 6 months postop and 12 months postop. Participants will also complete a series of standardized questionnaires at preop and 6 months, 12 months, and 24 month postop.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) is recognized as a highly effective procedure for alleviating pain and restoring function in patients with knee arthritis. Despite its high success rate, approximately 20% of patients remain dissatisfied with the outcomes, primarily due to loss of functional outcomes, persistent pain, and reduced knee range of motion. This has sparked a debate on the optimal surgical alignment technique in TKA-whether mechanical alignment (MA), or personalized alignment philosophies such as kinematic alignment (KA) or restricted kinematic alignment (rKA) provides superior patient outcomes.

MA traditionally targets a neutral 180-degree hip-knee-ankle (HKA) axis, as it was taught traditionally that this approach focuses on the longevity and stability of the implant. However, this one-size-fits-all philosophy overlooks individual anatomical differences. Personalized alignments such as KA customize the placement of prosthetic components to replicate each patient's unique knee geometry and ligament tensions. Personalized alignment philosophies aim to achieve a more natural knee motion, which may enhance patient satisfaction. The precision provided by robotic-assisted surgery has increasingly facilitated the implementation of personalized alignment philosophies in TKA. Recent evidence suggests that while MA and KA yield comparable outcomes in terms of knee functionality and motion, KA may improve satisfaction and the natural feel of the knee in certain groups, particularly those without severe preoperative deformities. There is also the emerging approach of restricted kinematic alignment (rKA) which aims to provide a compromise by aligning the prosthesis within safe anatomical limits, thus avoiding the extremes of anatomical variation. This approach tailors the surgery more closely to the individual's anatomy without the risks associated with the broader variances permitted in pure KA. Hypothetically, KA and rKA techniques should more closely replicate natural knee biomechanics and improve waking gait. There are advantages and disadvantages to these alignment philosophies which should be addressed with high-quality research. While there have been several previous randomized trials on MA vs KA and its variations, the evidence is still unclear with meta-analyses having conflicting findings.

Patients will be randomly assigned to either mechanical alignment or restricted kinematic alignment. All participants will receive robot-assisted TKA using the Stryker Mako surgical robot and Stryker implants. Perioperative care, postoperative pain medications, and rehabilitation will be standardized according to local standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 years or older
* Knee osteoarthritis requiring total knee arthroplasty
* Provide informed consent

Exclusion Criteria:

* Inability to provide informed consent (e.g. cognitive disability, language barrier)
* Revision knee surgery
* Simultaneous bilateral knee surgery
* Recent lower extremity surgery or trauma interfering with gait assessment
* A CT scan cannot be obtained prior to surgery
* Inability or unwillingness to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Gait Biomechanics | 12 months
  The primary outcome will be joint angles and walking characteristics (speed, step length, number of steps, consistency between sides) collected using an in-clinic markerless motion capture system. The system uses 10 synchronized optical cameras (60 Hz, Sony RXOII) placed strategically along the clinic hallways to maximize the viewing volume to capture patient movement characteristics. Advanced AI-driven software (Theia Markerless) is used to predict limb segment poses dynamically as the person moves through the space, and, combined with biomechanical modelling algorithms (Visual3D, C-Motion) can be used to accurately represent patient lower extremity 3D joint angles and other kinematic stride characteristics.

SECONDARY OUTCOMES:
Knee function | 24 months
  We will measure knee function using the Forgotten Joint Score (FJS-Knee). The FJS-Knee is a well validated and well-used 12 item questionnaire specifically used to measure function in elation to how natural a knee feels after total knee replacement surgery
Chronic post-surgical pain (CPSP) | 24 months
  We will use a modified version of the International Association for the Study of Pain's (IASP) definition of CPSP, to include a minimum threshold of pain severity: 1) Pain that developed after surgery; 2) Pain that lasts at least 3 months; 3) Other causes of pain have been excluded; 4) Pain caused by other conditions have been excluded; 5) Pain intensity at least 3/10 on a numeric rating score.
Quality of life | 24 months
  We will use the Euro-Qol 5 Dimensions-5L (EQ-5D-5L) questionnaire to assess health-related quality of life (HRQoL). The EQ-5D-5L is a well-validated and well-used quality of life instrument that can assess health utilities
Return to Function | 24 months
  We will use the Return To Function (RTF) questionnaire developed by Busse et al. at McMaster University. The RTF questionnaire is a 5 item questionnaire that has been used previously in orthopaedic trials to determine when a trial participant returns to work, leisure, and activities around the home after an injury or surgery

OTHER OUTCOMES:
Safety | 24 months
  We will collect all reoperations, serious adverse events (SAEs) and surgery-related non-serious AEs throughout the trial for safety monitoring purposes

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided